CLINICAL TRIAL: NCT07151014
Title: Prospective Single-center Study of a Cohort of Patients With Oral Lichen Planus: Cardiovascular and Prothrombotic Risk in Patients With Oral Lichen Planus (OLP).
Brief Title: Cardiovascular and Prothrombotic Risk in Patients With Oral Lichen Planus.
Acronym: LPO_RCP
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 7635
Record Dates: First submitted 2025-07-31; First posted 2025-09-02 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-10

CONDITIONS: Oral Lichen Planus
Keywords: oral lichen planus; Prothrombotic risk; trombophilia screening
MeSH Terms: conditions — Lichen Planus, Oral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: blood sample collection — blood sample collection in old patients in order to study the trombophilic risk

SUMMARY:
The primary objective is to evaluate the cardiovascular profile and the risk of thrombotic events in patients affected by Oral Lichen Planus.

DETAILED DESCRIPTION:
Evaluation of thrombophilia screening parameters, antiphospholipid antibody levels, and platelet aggregability in a cohort of patients affected by Oral Lichen Planus.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a clinical and histological diagnosis of Oral Lichen Planus
* Age > 18 years
* Patients who agree to sign the informed consent form

Exclusion Criteria:

* Patients under 18 years of age
* Patients who do not agree to sign the informed consent form
* Patients without a diagnosis of Oral Lichen Planus
* Patients with previously known cardiac diseases
* History of major cardiovascular events (myocardial infarction, ischemic stroke, TIA)
* Patients with overt heart failure (NYHA class III-IV)
* Cardiomyopathies not related to the studied risk factors (e.g., genetic hypertrophic cardiomyopathy)
* Patients undergoing anticoagulant therapy
* Patients with primary or secondary conditions associated with increased cardiovascular risk

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients affected by oral lichen planus
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-09-15 (Estimated); Study Completion 2027-02-15 (Estimated)

PRIMARY OUTCOMES:
Prothrombotic risk evaluation | From September 2025 to September 2026
  Primary Outcome Measure 1 Title: Prevalence of Natural Anticoagulant Deficiency
  * Description:
  Proportion of patients with Oral Lichen Planus (OLP) showing reduced functional activity of at least one natural anticoagulant (antithrombin III, protein C, or protein S) below the laboratory reference range, measured in plasma samples.
  * Time Frame:
  From September 2025 to September 2026
  * Unit of Measure:
  Percentage of participants with abnormal result (%). Primary Outcome Measure 2 Title: Prevalence of Antiphospholipid Antibody Positivity
  * Description:
  Proportion of OLP patients with positive antiphospholipid antibodies, defined as anticardiolipin IgG and/or IgM and/or anti-β2-glycoprotein I IgG/IgM above the laboratory cut-off, measured in serum.
  * Time Frame:
  From September 2025 to September 2026
  * Unit of Measure:
  Percentage of participants with abnormal result (%).

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-04-15): https://cdn.clinicaltrials.gov/large-docs/14/NCT07151014/Prot_SAP_000.pdf
  • Informed Consent Form (2025-04-15): https://cdn.clinicaltrials.gov/large-docs/14/NCT07151014/ICF_001.pdf